CLINICAL TRIAL: NCT01774396
Title: Clinical Trial On The Use Of Three Commercial Preparations Of Injectable Hyaluronic Acid (Emervel® Volume Lidocaine, Emervel® Deep Lidocaine And Emervel® Touch) In Hands Rejuvenation
Brief Title: Use Of Three Commercial Preparations Of Injectable Hyaluronic Acid In Hands Rejuvenation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-2012
Record Dates: First submitted 2012-12-28; First posted 2013-01-24 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Injuries to the Wrist and Hand
Keywords: Hands Rejuvenation, fillers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 2 (Other): The intervention will be the injection of Emervel® Volume Lidocaine alone in the dorsa of one hand and Emervel® Deep Lidocaine alone in the dorsa of the contralateral hand.
  Interventions: Drug: Emervel® Volume Lidocaine and Emervel® Deep Lidocaine
- group 1 (Experimental): EThe intervention will be the injection of mervel® Volume Lidocaine plus Emervel® Touch in the dorsa of one hand and Emervel® Deep Lidocaine plus Emervel® Touch in the dorsa of the contralateral hand
  Interventions: Drug: Emervel® Touch; Drug: Emervel® Volume Lidocaine and Emervel® Deep Lidocaine

INTERVENTIONS:
Drug: Emervel® Touch — Emervel® Touch will be injected only in the intervention group.
  Arms: group 1
Drug: Emervel® Volume Lidocaine and Emervel® Deep Lidocaine — Emervel® Volume Lidocaine and Emervel® Deep Lidocaine will be injected in the group #2.

SUMMARY:
Assessment of efficacy of hyaluronic acid - Emervel® Volume Lidocaine combined or not with Emervel® Touch and Emervel® Deep Lidocaine combined or not with Emervel® Touch in female patients with loss of fatty tissue in hands.

DETAILED DESCRIPTION:
This is a single center, phase IV, randomized, investigator-blind study of three different hyaluronic dermal filler injections for volume enhancing in the dorsum of the hands. As an investigator-blind study, only the investigators are unaware of which dermal fillers were injected in the dorsum of each hand.

ELIGIBILITY:
Inclusion Criteria:

* Subjects agreeing to take part of all procedures of the study (including pre-test, filler injection, photographs, etc.), after being fully informed on the objectives and nature of the investigations;
* Written Informed Consent;
* Treatment-naive patients for fillers in hands;
* Subjects of both genders over 18 years;
* Fitzpatrick skin phototypes I to VI;
* Subjects presenting a similar loss of fatty tissue on both hands, at least of 2 according the Validated Hand Grading Scale2;
* Medical history and physical examination which, based on the investigator's opinion, do not prevent the patient from taking part in the study and use the product under investigation;
* Female subjects of childbearing age should present a negative urine pregnancy test and should be using an effective contraceptive method;
* Availability of the subject throughout the duration of the study (208 days);
* Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol.

Exclusion Criteria:

* Pregnant women or women intending to become pregnant in the next 18 months;
* Subjects with known hypersensitivity to any hyaluronic acid products;
* Subjects with history of adverse effects, such as sensitivity to the components of the formula, or any other adverse effect, which in the investigator's opinion should prevent the patient from participating in the study;
* Subjects participating in other clinical trials;
* Any prior surgery or side effects at the hands area, or any prior cosmetic procedures, including permanent fillers, that may interfere with the results;
* Subjects with active inflammation or infection in the area to be treated;
* Subjects with a history of medical treatment non-adherence or showing unwillingness to adhere to the study protocol;
* Subjects presenting diseases such as coagulation disorders or under the use of anticoagulants, or any condition that, in the opinion of the investigator, can compromise the evaluation of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of hyaluronic acid - Emervel® Volume Lidocaine combined or not with Emervel® Touchand Emervel® Deep Lidocaine combined or not with Emervel® Touch in subjects with with loss of fatty tissue | at baseline and up to 180 days
  Assessment of efficacy of hyaluronic acid - Emervel® Volume Lidocaine combined or not with Emervel® Touch (Galderma) and Emervel® Deep Lidocaine combined or not with Emervel® Touch (Galderma) in female patients with loss of fatty tissue as a sign of aging on hands by Global Aesthetic Improvement scale1 and Hand Grading Scale2.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hexsel, MD, Principal Investigator — BRAZILIAN CENTER FOR STUDIES IN DERMATOLOGY
Locations (1):
- Brazilian center of Dermatology Studies, Porto Alegre, Rio Grande do Sul, Brazil